CLINICAL TRIAL: NCT03729245
Title: A Phase 3 Randomized Open Label Study to Compare NKTR-214 Combined With Nivolumab to the Investigator's Choice of Sunitinib or Cabozantinib in Patients With Previously Untreated Advanced Renal Cell Carcinoma
Brief Title: A Study of Bempegaldesleukin (NKTR-214: BEMPEG) in Combination With Nivolumab Compared With the Investigator's Choice of a Tyrosine Kinase Inhibitor (TKI) Therapy (Either Sunitinib or Cabozantinib Monotherapy) for Advanced Metastatic Renal Cell Carcinoma (RCC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-214-09; CA045002 (Other: Bristol-Myers Squibb Protocol ID)
Record Dates: First submitted 2018-10-29; First posted 2018-11-02 (Actual); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma
Keywords: Kidney Cancer; Kidney Neoplasms; Renal Cancer; Renal Neoplasms; CD122; CD122-Biased Agonist; CD122-Biased Cytokine; IL-2 receptor agonist; Immuno-oncology therapy; NKTR-214; Nivolumab; Opdivo®; PD-L1; PD-1; Bempegaldesleukin; IL-2; BEMPEG; CD122-Preferential; IL-2 pathway agonist; Checkpoint inhibition; Immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — bempegaldesleukin; Sunitinib; Nivolumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination of bempegaldesleukin + nivolumab (Experimental): Patients in Arm A will receive bempegaldesleukin in combination with nivolumab.
  Interventions: Biological: bempegaldesleukin; Biological: nivolumab
- sunitinib or cabozantinib (Active Comparator): Patients in Arm B will receive the Investigator's choice of either one of two treatment options.
  Interventions: Drug: sunitinib; Drug: cabozantinib

INTERVENTIONS:
Biological: bempegaldesleukin — Specified dose on specified days
  Other Names: BEMPEG; BMS-986321
  Arms: Combination of bempegaldesleukin + nivolumab
Drug: sunitinib — Specified dose on specified days
  Other Names: Sutent®
  Arms: sunitinib or cabozantinib
Biological: nivolumab — Specified dose on specified days
  Other Names: Opdivo®; BMS-936558
  Arms: Combination of bempegaldesleukin + nivolumab
Drug: cabozantinib — Specified dose on specified days
  Other Names: Cabometyx®
  Arms: sunitinib or cabozantinib

SUMMARY:
The main purpose of this study is to compare the objective response rate (ORR) and overall survival (OS) of bempegaldesleukin (NKTR-214: BEMPEG) combined with nivolumab to that of tyrosine kinase inhibitor (TKI) monotherapy (sunitinib or cabozantinib) in IMDC intermediate- or poor-risk patients and IMDC all-risk patients with previously untreated advanced renal cell carcinoma (RCC).

ELIGIBILITY:
Key Inclusion Criteria:

* Provide written, informed consent to participate in the study and follow the study procedures
* Karnofsky Performance Status (KPS) of at least 70%
* Measurable disease per mRECIST 1.1 criteria
* Histologically confirmed RCC with a clear-cell component (may have sarcomatoid features); advanced (not amenable to curative surgery or radiation therapy) or metastatic (AJCC Stage IV) RCC
* Patients with any International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) score (favorable-, intermediate-, or poor-risk) are eligible. At least one IMDC prognostic factor must be present to qualify as either intermediate- or poor-risk renal cell carcinoma.
* No prior systemic therapy (including neoadjuvant, adjuvant, or vaccine therapy) for RCC

Key Exclusion Criteria:

* An active, known or suspected autoimmune disease that has required systemic treatment within the past 3 months (exceptions exist)
* Patients who have a known additional malignancy that is progressing or requires active treatment (exceptions exist)
* Any tumor invading the wall of a major blood vessels
* Any tumor invading the gastrointestinal (GI) tract or any evidence of endotracheal or endobronchial tumor within 28 days prior to randomization
* Need for >2 medications for management of hypertension (including diuretics)
* History of pulmonary embolism, deep vein thrombosis (not including tumor thrombus), or clinically significant thromboembolic event within 3 months of randomization

Additional protocol defined inclusion/exclusion criteria and exceptions apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (95):
- United States (20):
  - Alaska Urological, Anchorage, Alaska
  - Western Regional Medical Center - CTCA - PPDS, Goodyear, Arizona
  - CARTI Cancer Center, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - University of California Irvine, Orange, California
  - Innovative Clinical Research Institute, Whittier, California
  - University of Miami, Miami, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - North Shore Hematology Oncology Association PC, Port Jefferson Station, New York
  - Kettering Medical Center, Kettering, Ohio
  - Providence Cancer Institute, Franz Clinic, Portland, Oregon
  - Lehigh Valley Physician Group (LVPG) - Hematology Oncology, Allentown, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center - CTCA, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Hospital - PPDS, Salt Lake City, Utah
- Argentina (11):
  - Centro de Investigación Clínica - Clínica Viedma, Viedma, Río Negro Province
  - Centro de Investigación Pergamino S.A, Buenos Aires
  - Centro Médico Austral, Buenos Aires
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires
  - Centro Médico Privado CEMAIC, Córdoba
  - Sanatorio Allende S.A., Córdoba
  - Sanatorio Privado Duarte Quirós, de Clínica Colombo S.A., Córdoba
  - Centro Oncologico Riojano Integral (cori), La Rioja
  - Hospital Provincial Del Centenario, Rosario
  - CAIPO Centro para la atención integral del paciente oncológico, San Miguel de Tucumán
  - Sanatorio Parque de Rosario, Santa Fe
- Australia (5):
  - Orange Cancer Centre, Orange, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Barwon Health, Parkville, Victoria
- Brazil (27):
  - Centro de Oncologia Da Bahia, Salvador, Estado de Bahia
  - Ensino E Terapia de Inovação Clínica Assistência Multidiciplinar Em Oncologia Ética, Salvador, Estado de Bahia
  - Cenantron - Centro Avancado de Tratamento Oncologico Ltda, Belo Horizonte, Minas Gerais
  - Oncocentro, Belo Horizonte, Belo Horizonte, Minas Gerais
  - Liga Paranaense de Combate Ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - Liga Norte Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Associação Hospital de Caridade Ijuí, Ijuí, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Universidade Federal do Rio Grande do Sul - UFRGS, Porto Alegre, Rio Grande do Sul
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Clínica de Oncologia de Porto Alegre SS Ltda, Rio Grande, Rio Grande do Sul
  - Instituto Joinvilense de Hematologia E Oncologia, Joinville, Santa Catarina
  - Fundação Pio XII Hospital de Câncer de Barretos, Barretos, São Paulo
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Fundação do ABC - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Instituto de Pesquisas Clínicas Para Estudos Multicêntricos, Caxias do Sul
  - Instituto Do Câncer Do Ceará ICC, Fortaleza
  - Animi, Lages
  - Instituto Nacional de Câncer, Rio de Janeiro
  - Instituto COI de Pesquisa, Educação e Gestão, Rio de Janeiro
  - Hospital de Base Da Faculdade de Medicina de São José Do Rio Preto, São José do Rio Preto
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Fundação Antônio Prudente - AC Camargo Câncer Center, São Paulo
  - Hospital Santa Marcelina, São Paulo
- Chile (8):
  - Corporacion de Beneficencia Osorno, Osorno, Los Lagos Region
  - Clinical Research Chile SpA, Valdivia, Los Ríos Region
  - Oncovida, Santiago
  - Clinica Santa Maria, Santiago
  - Fundación Arturo López Pérez (FALP) - PPDS, Santiago
  - Centro Investigacion Clinica Del Sur, Temuco
  - Oncocentro APYS, Viña del Mar
  - Centro de Investigaciones Clínicas Vina del Mar, Viña del Mar
- Mexico (5):
  - Health Pharma Professional Research S.A de C.V., Mexico City, Mexico City
  - Centro de Investigacion Clinica Chapultepec S.A. de C.V., Morelia, Michoacán
  - Axis Heilsa S. De R.L. de C.V., Monterrey, Nuevo León
  - Accelerium, S. de R.L. de C.V., Monterrey
  - Unidad Médica Onco-Hematológica, Puebla City
- Auckland City Hospital, Auckland, New Zealand
- Peru (4):
  - Clinica Peruana Americana, Trujillo, La Lobertad
  - Clinica Internacional S.A. - Sede San Borja, Lima
  - ONCOCARE S.A.C. (Clinica Aliada), Lima
  - Hospital Nacional Cayetano Heredia, Lima
- Russia (12):
  - Altay Regional Oncology Center, Barnaul
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk
  - LLC Evimed, Chelyabinsk
  - Kursk Regional Oncology Centre, Kursk
  - Central Clinical Hospital With Polyclinic of President Administration of RF, Moscow
  - Federal State Institution Medical Radiology Research Center, Obninsk
  - Clinical Oncology Dispensary, Omsk
  - PMI Euromedservice, Pushkin
  - Hospital Orkli LLC, Saint Petersburg
  - Railway Clinical Hospital JSC RZhD, Saint Petersburg
  - State Institution of Healthcare "Volgograd Regional Urology and Nephrology Centre", Volzhskiy
  - Regional Clinical Oncology Hospital, Yaroslavl
- Singapore (2):
  - National Cancer Centre, Singapore
  - Oncocare Cancer Centre, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tannir NM, Formiga MN, Penkov K, Kislov N, Vasiliev A, Gunnar Skare N, Hong W, Dai S, Tang L, Qureshi A, Zalevsky J, Tagliaferri MA, George D, Agarwal N, Pal S. Bempegaldesleukin Plus Nivolumab Versus Sunitinib or Cabozantinib in Previously Untreated Advanced Clear Cell Renal Cell Carcinoma: A Phase III Randomized Study (PIVOT-09). J Clin Oncol. 2024 Aug 10;42(23):2800-2811. doi: 10.1200/JCO.23.02082. Epub 2024 Jun 5. PMID 38838287

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination of Bempegaldesleukin + Nivolumab: Patients in Arm A will receive bempegaldesleukin in combination with nivolumab.
  Bempegaldesleukin (NKTR-214) 0.006 mg/kg intravenous (IV) every 3 weeks (q3w) combined with nivolumab 360 mg IV q3w
- Sunitinib or Cabozantinib: Patients in Arm B will receive the Investigator's choice of either one of two treatment options.
  Sunitinib 50 mg per orally (po) once daily for 4 weeks followed by 2 weeks off OR Cabozantinib 60 mg po once daily
Period: Overall Study
Arm/Group | Combination of Bempegaldesleukin + Nivolumab | Sunitinib or Cabozantinib
Started | 311 | 312
Completed | 289 | 287
Not Completed | 22 | 25
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 16 | 19
Not completed — Patient did not complete the end of study form but is not followed on the study anymore. | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total of 623 patients were randomized in the ITT International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) All-risk population, including 514 patients for the ITT I/P-risk population:
  * NKTR-214/nivolumab: 311 and 256, respectively
  * Sunitinib or cabozantinib: 312 and 258, respectively
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination of Bempegaldesleukin + Nivolumab | Sunitinib or Cabozantinib | Total
Number analyzed (Participants) | 311 | 312 | 623
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (9.74) | 60.8 (10.24) | 61.2 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 80 | 155
  Male | 236 | 232 | 468
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 148 | 131 | 279
  Not Hispanic or Latino | 157 | 172 | 329
  Unknown or Not Reported | 6 | 9 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 271 | 272 | 543
  Black or African American | 7 | 6 | 13
  Asian | 5 | 7 | 12
  American Indian or Alaska Native | 14 | 8 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Not Reported | 7 | 8 | 15
  Other | 7 | 11 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 49 | 28 | 77
  Singapore | 3 | 2 | 5
  United States | 41 | 50 | 91
  Russia | 95 | 108 | 203
  New Zealand | 4 | 2 | 6
  Brazil | 68 | 82 | 150
  Mexico | 16 | 11 | 27
  Australia | 7 | 8 | 15
  Chile | 19 | 16 | 35
  Peru | 9 | 5 | 14
Karnofsky Performance Status (KPS) Score [Number; unit: participants] — The Karnofsky Performance Status (KPS) scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities; For example: Score of 100 = Normal, no complaints, no evidence of disease. 80 = Normal activity with effort; some signs or symptoms of disease. 50 = Requires considerable assistance and frequent medical care. 30 = Severely disabled, hospitalization indicated. Death not imminent. 0 = Dead
  participants
    KPS < 80 | 77 | 75 | 152
    KPS >= 80 | 234 | 237 | 471

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per mRECIST 1.1 by BICR in IMDC All-risk Patients and Intermediate- or Poor (I/P)-Risk Patients With Previously Untreated Advanced RCC
Description: ORR using modified Response Evaluation Criteria in Solid Tumors (mRECIST) 1.1 by Blinded Independent Central Review (BICR) in International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) All-risk patients and intermediate- or poor-risk patients.
  ORR is defined as the proportion of enrolled participants who achieved a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR is calculated as the sum of CR and PR.
Time Frame: Approximately 32 months
Population: A total of 623 patients randomized in the ITT All-risk population, including 514 patients for the ITT I/P-risk population:
  * NKTR-214/nivolumab: 311 (ITT All-risk population) and 256 (ITT I/P-risk population), respectively
  * Sunitinib or Cabozantinib (TKI): 312 (ITT All-risk population) and 258 (ITT I/P-risk population), respectively
Measure: Count of Participants; unit: Participants
Arm/Group | Combination of Bempegaldesleukin + Nivolumab | Sunitinib or Cabozantinib
Number analyzed (Participants) | 311 | 312
Participants
  ORR per mRECIST 1.1 by BICR, ITT All-risk population | 73 | 109
  ORR per mRECIST 1.1 by BICR, ITT I/P-risk population: number analyzed (Participants) | 256 | 258
  ORR per mRECIST 1.1 by BICR, ITT I/P-risk population | 59 | 79

2. Primary Outcome: Overall Survival (OS) in IMDC All-Risk and Intermediate- or Poor-risk Patients With Previously Untreated Advanced RCC
Description: OS is defined as the time from date of first dose to the date of death from any cause. Patients without a date of death were censored at their last known alive date.
Time Frame: Approximately 32 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination of Bempegaldesleukin + Nivolumab | Sunitinib or Cabozantinib
Number analyzed (Participants) | 311 | 312
months
  OS, ITT All-risk population | NA [29.0 to NA] — Median and upper CI was not estimable due to insufficient number of events. | NA [NA to NA] — Median and 95% CI was not estimable due to insufficient number of events.
  OS, ITT I/P-risk population: number analyzed (Participants) | 256 | 258
  OS, ITT I/P-risk population | 29 [25.6 to NA] — Upper CI was not estimable due to insufficient number of events. | NA [25.6 to NA] — Median and upper CI was not estimable due to insufficient number of events.

3. Secondary Outcome: Progression Free Survival (PFS) Per mRECIST 1.1 by BICR in IMDC All-risk Patients and Intermediate- or Poor (I/P)-Risk Patients With Previously Untreated Advanced RCC
Description: Progression-free survival is defined as the time between the date of randomization and the first date of documented tumor progression using mRECIST 1.1 per BICR or death due to any cause, whichever comes first.
Time Frame: Approximately 32 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combination of Bempegaldesleukin + Nivolumab | Sunitinib or Cabozantinib
Number analyzed (Participants) | 311 | 312
Months
  PFS per mRECIST 1.1. by BICR, ITT All-risk population | 8.2 [6.2 to 10.0] | 10.3 [8.5 to 12.4]
  PFS per mRECIST 1.1. by BICR, ITT I/P-risk population: number analyzed (Participants) | 256 | 258
  PFS per mRECIST 1.1. by BICR, ITT I/P-risk population | 6.4 [4.6 to 8.3] | 9.2 [8.3 to 12.2]

ADVERSE EVENTS:
Time Frame: AEs will be reported starting immediately after the patient has been administered the first dose of study drug(s) until 100 days after the last dose of all study drug(s), up to 38 months. All ongoing non-serious AEs will be followed until resolution, the patient is lost to follow-up, patient death, or until the last Safety Follow-Up Visit. If the AE has not completely resolved by the last Safety Follow-Up Visit, the final outcome of these ongoing AEs will be captured.
Arm/Group | Combination of Bempegaldesleukin + Nivolumab | Sunitinib or Cabozantinib
All-Cause Mortality (participants affected / at risk) | 109/310 | 114/306
Serious Adverse Events (participants affected / at risk) | 113/310 | 91/306
Other Adverse Events (participants affected / at risk) | 307/310 | 304/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Bempegaldesleukin + Nivolumab (N=310) | Sunitinib or Cabozantinib (N=306)
Corona virus infection (Infections and infestations) | 13 | 3
Pneumonia (Infections and infestations) | 9 | 2
Pneumonia viral (Infections and infestations) | 4 | 2
Sepsis (Infections and infestations) | 4 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Infection (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endotoxic shock (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Parotid abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tonsillitis bacterial (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 2 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 4 | 1
Seizure (Nervous system disorders) | 3 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 3
Syncope (Nervous system disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 2
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Conus medullaris syndrome (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0
Sensory loss (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2
Acute coronary syndrome (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 5
Haematuria (Renal and urinary disorders) | 0 | 3
Renal impairment (Renal and urinary disorders) | 1 | 2
Anuria (Renal and urinary disorders) | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 7 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 2
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Generalised oedema (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 1
Asthenia (General disorders) | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Contrast media reaction (Immune system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0
Genital ulceration (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Bempegaldesleukin + Nivolumab (N=310) | Sunitinib or Cabozantinib (N=306)
Diarrhoea (Gastrointestinal disorders) | 87 | 161
Nausea (Gastrointestinal disorders) | 100 | 119
Vomiting (Gastrointestinal disorders) | 61 | 74
Abdominal pain (Gastrointestinal disorders) | 32 | 50
Constipation (Gastrointestinal disorders) | 30 | 49
Stomatitis (Gastrointestinal disorders) | 9 | 64
Abdominal pain upper (Gastrointestinal disorders) | 21 | 34
Dyspepsia (Gastrointestinal disorders) | 14 | 35
Dry mouth (Gastrointestinal disorders) | 15 | 17
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 16
Fatigue (General disorders) | 72 | 87
Pyrexia (General disorders) | 121 | 28
Asthenia (General disorders) | 77 | 57
Oedema peripheral (General disorders) | 36 | 39
Chills (General disorders) | 45 | 27
Influenza like illness (General disorders) | 51 | 8
Mucosal inflammation (General disorders) | 8 | 39
Non-cardiac chest pain (General disorders) | 17 | 18
Face oedema (General disorders) | 17 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 105 | 33
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 113
Rash (Skin and subcutaneous tissue disorders) | 74 | 28
Pruritus generalised (Skin and subcutaneous tissue disorders) | 53 | 18
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 33
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 | 13
Erythema (Skin and subcutaneous tissue disorders) | 24 | 6
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 27
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 16
Aspartate aminotransferase increased (Investigations) | 17 | 71
Alanine aminotransferase increased (Investigations) | 22 | 65
Blood creatinine increased (Investigations) | 48 | 37
Weight decreased (Investigations) | 28 | 56
Lipase increased (Investigations) | 28 | 44
Amylase increased (Investigations) | 14 | 40
Blood alkaline phosphatase increased (Investigations) | 15 | 30
Blood thyroid stimulating hormone increased (Investigations) | 11 | 33
Platelet count decreased (Investigations) | 1 | 41
Blood creatine phosphokinase increased (Investigations) | 8 | 28
Body temperature increased (Investigations) | 34 | 1
Blood lactate dehydrogenase increased (Investigations) | 6 | 28
Blood pressure increased (Investigations) | 4 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 90 | 76
Back pain (Musculoskeletal and connective tissue disorders) | 53 | 57
Myalgia (Musculoskeletal and connective tissue disorders) | 70 | 38
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 31
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 | 16
Decreased appetite (Metabolism and nutrition disorders) | 82 | 103
Hyperkalaemia (Metabolism and nutrition disorders) | 21 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 21
Hyponatraemia (Metabolism and nutrition disorders) | 13 | 22
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 17
Anaemia (Blood and lymphatic system disorders) | 57 | 109
Neutropenia (Blood and lymphatic system disorders) | 19 | 86
Eosinophilia (Blood and lymphatic system disorders) | 82 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 73
Leukopenia (Blood and lymphatic system disorders) | 3 | 41
Lymphopenia (Blood and lymphatic system disorders) | 5 | 18
Headache (Nervous system disorders) | 87 | 90
Dizziness (Nervous system disorders) | 52 | 40
Dysgeusia (Nervous system disorders) | 18 | 65
Hypotonia (Nervous system disorders) | 16 | 1
Hypothyroidism (Endocrine disorders) | 74 | 129
Hyperthyroidism (Endocrine disorders) | 45 | 17
Corona virus infection (Infections and infestations) | 36 | 37
Urinary tract infection (Infections and infestations) | 14 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 54 | 43
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 | 24
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 17
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17 | 2
Hypertension (Vascular disorders) | 29 | 112
Hypotension (Vascular disorders) | 43 | 7
Insomnia (Psychiatric disorders) | 34 | 49
Anxiety (Psychiatric disorders) | 26 | 31
Chronic kidney disease (Renal and urinary disorders) | 15 | 18
Proteinuria (Renal and urinary disorders) | 2 | 31
Infusion related reaction (Injury, poisoning and procedural complications) | 18 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT03729245/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT03729245/SAP_001.pdf